CLINICAL TRIAL: NCT02110238
Title: Multicenter, Randomized, Double-Blind, Parallel Controlled Non-Inferiority Clinical Trial Comparing 3 Weekly Intra-articular Injections of SUPARTZ® vs 3 Weekly Intra-articular Injections of Euflexxa® for Treatment of Knee OA
Brief Title: Non-Inferiority Study Comparing 3 Weekly Injections of SUPARTZ® vs 3 Weekly Injections of Euflexxa® for Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioventus LLC (Industry)
Collaborators: Seikagaku Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13SUP301
Record Dates: First submitted 2014-04-03; First posted 2014-04-10 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee pain; Supartz; Euflexxa; HA; hyaluronic acid
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Euflexxa (Active Comparator): Euflexxa® (hyaluronic acid of bacterial origin)
  Interventions: Device: Euflexxa
- Supartz (Experimental): SUPARTZ® (hyaluronic acid of avian origin)
  Interventions: Device: Supartz

INTERVENTIONS:
Device: Supartz — Treatment is 3 injections over 2 weeks; Week 0 (baseline), Week 1, and Week 2.
  Arms: Supartz
Device: Euflexxa — Treatment is 3 injections over 2 weeks; Week 0 (baseline), Week 1, and Week 2.
  Arms: Euflexxa

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of three weekly intra-articular injections of SUPARTZ to three weekly intra-articular injections of Euflexxa for the relief of knee OA.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate non-inferiority of three weekly intra-articular injections of SUPARTZ to three weekly intra-articular injections of Euflexxa for the relief of knee joint pain in subjects with osteoarthritis (OA) of the knee as measured by the VAS (0-100 mm) Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain subscale score Change from Baseline (CFB) over Weeks 3, 6, 12.

Safety will be accessed by recording adverse events, concomitant medications, physical examinations, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of symptomatic osteoarthritis of the study knee as classified according to Altman criteria.
* Symptoms in study knee for at least one year prior to the screening visit
* Verified OA of the study knee of Grade 2 or 3 according to a modification of the grading system of Kellgren-Lawrence (K-L) radiographic severity.
* Willingness to discontinue NSAIDs (systemic and topical) and non-acetaminophen analgesic use seven days or five half-lives prior to the first injection and throughout the study.

Exclusion Criteria:

* Inability to perform a 50 foot walk test.
* Subjects with rheumatoid arthritis, joint infection, other inflammatory and metabolic arthritis, Lupus or dermatologic disorder or skin conditions in close proximity to study knee that would preclude safe intra-articular injections.
* Prior hyaluronic acid injections into the study knee within six months of the screening visit.
* Intra-articular or intra-muscular steroid injections within three months of the screening visit or during study participation. Oral corticosteroids within four weeks of the screening visit or during study participation.
* History of surgical treatment to the study knee or arthroscopic intervention within three months prior to the screening visit.
* Clinically apparent tense effusion of the study knee on examination determined by either a positive bulge sign or positive ballottement of the patella (patellar tap).
* Subjects with clinically diagnosed symptomatic OA of the hip.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Strand, MD, Principal Investigator — Stanford University
Locations (1):
- Triangle Orthopaedic Associates, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 outpatient medical clinics enrolled subjects over 4.5 months
Period: 12 Week Pivotal Phase
Arm/Group | Euflexxa | Supartz
Started | 212 (One subject was randomized but not treated. As a result there were 211 safety subjects) | 209
Completed | 202 | 200
Not Completed | 10 | 9
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3
Period: 14 Week Blinded Extension Phase
Arm/Group | Euflexxa | Supartz
Started | 202 | 200
Completed | 190 | 188
Not Completed | 12 | 12
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 2 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: All but 1 subject who discontinued after being randomized to Euflexxa but unable to tolerate the injection procedure. This subject did not receive any of the study device via injection.
Groups:
- Euflexxa: Euflexxa® Treatment is 3 injections over 2 weeks; Week 0 (baseline), Week 1, and Week 2.
- Supartz: SUPARTZ® Treatment is 3 injections over 2 weeks; Week 0 (baseline), Week 1, and Week 2.
- Total: Total of all reporting groups
Arm/Group | Euflexxa | Supartz | Total
Number analyzed (Participants) | 211 | 209 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.33) | 59.3 (9.30) | 60.1 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 138 | 273
  Male | 76 | 71 | 147

OUTCOME MEASURES:

1. Primary Outcome: WOMAC VAS (0:None -100:Extreme) Pain Subscale Score Change From Baseline
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) 0-100mm Pain subscale score Change from Baseline (CFB). Over weeks 3, 6, and 12 least square mean difference in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Visual Analog Scale (VAS) (0mm:None - 100mm:Extreme) pain subscale score Change from Baseline (CFB). A single estimate of least squares mean was calculated using data from baseline, weeks 3, 6, and 12.
Time Frame: Change from Baseline (CFB) over Weeks 3, 6, and 12
Population: Per Protocol: All subjects with at least 1 post baseline primary outcome measure and no important protocol deviations.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter
Arm/Group | Euflexxa | Supartz
Number analyzed (Participants) | 189 | 195
millimeter | 30.15 [27.59 to 32.71] | 26.85 [24.35 to 29.35]
Statistical Analysis 1: Comparison: Euflexxa vs Supartz; Test type: Non-Inferiority or Equivalence — A VAS (0-100 mm) WOMAC Pain subscale score CFB; an equal n t-test for non-inferiority of means; a non-inferiority margin of -8 mm; change standard deviation of 26 mm; two-sided alpha=0.05; 80% power; an expected mean difference of 0, and a drop-out plus important deviation percentage of approximately 20% were used to establish study sample size; Least square mean difference = -3.30, 95% CI 2-sided [-6.77 to 0.17] — A MERM regression model was fit to the change from baseline at weeks 3, 6, and 12. The over weeks 3, 6, and 12 "single point estimate" least square mean change was calculated for both arms, the difference and its 95% confidence interval calculated

ADVERSE EVENTS:
Time Frame: 26 Weeks (12 week primary period plus 14 week extension phase)
Groups:
- Euflexxa: Euflexxa® (hyaluronic acid of bacterial origin) Treatment is 3 injections over 2 weeks; Week 0 (baseline), Week 1, and Week 2.
- Supartz: SUPARTZ® (hyaluronic acid of avian origin) Treatment is 3 injections over 2 weeks; Week 0 (baseline), Week 1, and Week 2.
Arm/Group | Euflexxa | Supartz
Serious Adverse Events (participants affected / at risk) | 6/211 | 1/209
Other Adverse Events (participants affected / at risk) | 59/211 | 60/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Euflexxa (N=211) | Supartz (N=209)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax tramatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Euflexxa (N=211) | Supartz (N=209)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 15
Headache (Nervous system disorders) | 25 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No